CLINICAL TRIAL: NCT04777708
Title: Pilot Feasibility Study of Intratumoral BO-112 in Combination With Pembrolizumab for Advanced Hepatocellular Carcinoma
Brief Title: BO-112 and Pembrolizumab for the Treatment of PD-1/PD-L1 Refractory Liver Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Withdrawn by sponsor
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Highlight Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-000276; NCI-2021-00994 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-000276 (Other: UCLA / Jonsson Comprehensive Cancer Center)
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Advanced Hepatocellular Carcinoma; BCLC Stage B Hepatocellular Carcinoma; BCLC Stage C Hepatocellular Carcinoma; Refractory Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — BO-112; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (pembrolizumab, BO-112) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 of odd number cycles. Patients also receive BO-112 by intratumoral injection on day 1, 8, and 15 of cycle 1, and day 15 of subsequent cycles. Treatment repeats every 3 weeks for up to 17 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nanoplexed Poly I:C BO-112; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Nanoplexed Poly I:C BO-112 — Given by intratumoral injection
  Other Names: BO 112; BO-112; BO112; Nanoplexed Poly IC BO-112; Nanoplexed Polyinosinic:Polycytidylic Acid BO-112
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This early phase I trial evaluates the side effects of BO-112 and pembrolizumab and how well they work in treating patients with Barcelona Clinic Liver Cancer (BCLC) stage B or C liver cancer. Immunotherapy with BO-112, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the tumor, and may interfere with the ability of tumor cells to grow and spread. Giving BO-112 and pembrolizumab may help treat patients with liver cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the early efficacy and safety for the combination of intratumoral nanoplexed poly I:C BO-112 (BO-112) in combination with pembrolizumab in patients with advanced hepatocellular carcinoma (HCC) who have progressed on prior anti-PD-1/PD-L1 therapy.

SECONDARY OBJECTIVES:

I. To further elucidate efficacy endpoints of the combination the combination of BO-112 with pembrolizumab.

II. To demonstrate the efficacy of BO-112 from its hypothesized mechanism of action.

CORRELATIVE RESEARCH OBJECTIVES:

I. Peripheral blood will be collected to assess changes in circulating cluster of differentiation 4 (CD4+), cluster of differentiation 8 (CD8+), natural killer (NK), and dendritic cells.

II. Peripheral blood will be collected to assess leukocyte expression of interferon beta induced genes in conjunction with intratumoral studies to demonstrate increased intratumoral interferon beta and other hypothesized biomarkers.

III. A baseline biopsy will be collected on cycle 1 day 1 and at cycle 2 day 15 (done at the same time as intratumoral injection).

IIIa. From these biopsies, intratumoral CD4+, CD8+ expression and cluster of differentiation 56 (CD56+) expression (NK cells) will be measured by immunohistochemistry on the baseline biopsy and the biopsy on cycle 2 day 15.

IIIb. Myeloid dendritic cells will be assessed by flow cytometry, as their activity correlates with Toll-like receptor 3 (TLR3) activation.

IIIc. Percentage of cells with apoptosis and necrosis will be assessed. IIId. The tumor microenvironment will be assessed by ribonucleic acid (RNA) expression profiling with nCounter Pancancer Immune Profiling Panel given its extensive validation to date.

IV. To assess the potential of immune-related Response Evaluation Criteria in Solid Tumors (RECIST) (iRECIST) to determine disease control as compared to RECIST 1.1.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 of odd number cycles. Patients also receive BO-112 by intratumoral injection on day 1, 8, and 15 of cycle 1, and day 15 of subsequent cycles. Treatment repeats every 3 weeks for up to 17 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 8 weeks for 1 year, and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are at least 18 years of age on the day of signing informed consent with confirmed diagnosis of hepatocellular carcinoma by radiology, histology, or cytology (fibrolamellar and mixed hepatocellular/cholangiocarcinoma subtypes are not eligible) will be enrolled in this study.

  * Radiologic confirmation diagnosis is provided by the study site. Clinically confirmed diagnosis of HCC as per the American Association for the Study of Liver Diseases (AASLD) criteria, which requires:

    * Radiographically evident cirrhosis AND
    * A liver mass that shows arterial phase hyperenhancement on triphasic computed tomography (CT) or magnetic resonance imaging (MRI), AND EITHER:

      * Is >= 20 mm with either non-peripheral portal washout or an enhancing capsule OR
      * Is 10-19 mm with non-peripheral portal venous washout AND an enhancing capsule
* Have Barcelona Clinic Liver Cancer (BCLC) stage C disease, or BCLC stage B disease not amenable to locoregional therapy or refractory to locoregional therapy, and not amenable to a curative treatment approach
* Have a Child-Pugh class A liver score within 14 days of first dose of study drug
* Have a predicted life expectancy of > 3 months
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

  * Not a woman of childbearing potential (WOCBP) OR
  * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days/weeks (corresponding to time needed to eliminate any study treatment(s) after the last dose of study treatment.
  * Note: a male participant is not required to use contraception during the treatment period for pembrolizumab and BO-112. BO-112 does not have any evidence of genotoxicity at any dose
* Participants must have progressed radiographically on treatment with an anti-PD-1/L1 monoclonal antibody (mAb) administered either as monotherapy or in combination with other checkpoint inhibitors or other adjunct therapies. Participants must not have received BO-112 previously. PD-1/L1 treatment progression is defined by meeting all of the following criteria:

  * Has received at least 2 doses of an approved anti-PD-1/L1 mAb
  * Has demonstrated progressive disease after anti-PD-1/L1 as defined by RECIST version (v)1.1
  * Progressive disease has been documented within 12 weeks from the last dose of anti-PD-1/L1 mAb

    * Progressive disease is determined according to RECIST 1.1
    * This determination is made by the investigator. Once disease progression is confirmed, the initial date of disease progression documentation will be considered the date of disease progression
* The participant (or legally acceptable representative if applicable) provides written informed consent for the trial
* Have measurable disease based on RECIST 1.1 and accessible for intratumoral injection and biopsy. (This lesion to be injected cannot infiltrate the main hepatic vessels.) Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions after the administration of the radiotherapy
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to cycle 1 day 1 (C1D1)
* Subjects with chronic infection by hepatitis C virus (HCV) who are treated (successfully or treatment failure) or untreated are allowed on study. In addition, subjects with successful HCV treatment are allowed as long as there are >= 4 weeks between achieving sustained viral response (SVR12) and start of study drug.

  * Successful HCV treatment definition: SVR12
* Has been treated with anti-hepatitis B therapy. Controlled (treated) hepatitis B subjects will be allowed if they meet the following criteria:

  * Antiviral therapy for hepatitis B virus (HBV) must be given for at least 12 weeks and HBV viral load must be less than 100 IU/mL prior to first dose of study drug. Subjects on active HBV therapy with viral loads under 100 IU/mL should stay on the same therapy throughout study treatment
  * Subjects who are hepatitis B core antibody (anti-HBc) (+), negative for hepatitis B surface antigen (HBsAg), and negative or positive for hepatitis B surface antibody (anti-HBs), and who have an HBV viral load under 100 IU/mL, do not require HBV anti-viral prophylaxis
* Absolute neutrophil count (ANC) >= 1200/uL (microliters) (within 7 days prior to the start of study treatment)
* Platelets >= 60 000/uL (within 7 days prior to the start of study treatment)
* Hemoglobin >= 8.0 g/dL (within 7 days prior to the start of study treatment)

  * Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can be used in place of creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN (within 7 days prior to the start of study treatment)

  * Creatinine clearance (CrCl) should be calculated per institutional standard
* Total bilirubin =< 3 mg/dL, or direct bilirubin =< ULN for those with total bilirubin > 2 mg/dL (within 7 days prior to the start of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 5 x ULN (within 7 days prior to the start of study treatment)
* Albumin >= 2.8 g/dL (within 7 days prior to the start of study treatment)

  * Note: No albumin supplement (or BCAA) allowed within the last 14 days
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.7 unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants (within 7 days prior to the start of study treatment)
* Activated partial thromboplastin time (aPTT) =< 1.7 unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants (within 7 days prior to the start of study treatment)

Exclusion Criteria:

* A WOCBP who has a positive urine pregnancy test within 72 hours prior to C1D1. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note: in the event that 72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication
* Has received prior systemic anti-cancer therapy including investigational agents within 4 weeks prior to C1D1. Note: Participants must have recovered from all adverse events (AEs) due to previous therapies to=< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment
* Has had esophageal or gastric variceal bleeding within the last 6 months
* Has clinically apparent ascites on physical examination

  * Note: ascites detectable on imaging studies only are allowed
* Has had clinically diagnosed hepatic encephalopathy in the last 3 months. Subjects on rifaximin or lactulose to control their hepatic encephalopathy are not allowed
* Has received locoregional therapy to liver (transcatheter chemoembolization [TACE], transcatheter embolization [TAE], hepatic arterial infusion [HAI], radiation, radioembolization, or ablation) within 4 weeks prior to the first dose of study drug. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-liver, non-central nervous system (CNS) disease
* Prior treatment with any Toll-like receptor (TLR) agonist
* Has liver lesions with macroscopic tumor infiltration into the main portal vein, hepatic vein, or inferior vena cava
* Has had major surgery to liver or other site within 4 weeks prior to the first dose of study drug
* Has had a minor surgery (i.e., simple excision, tooth extraction) =< 7 days prior to the first dose of study treatment (cycle 1, day 1)
* Contraindications to tumor biopsy and injections of the hepatic metastasis(es), such as coagulopathy, therapeutic dose anticoagulant treatment and/or treatment with long-acting agents such as clopidogrel which cannot be safely stopped
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed
* Has a history of a second malignancy, unless potentially curative treatment has been completed with no evidence of malignancy for 1 year. Note: The time requirement does not apply to participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, in situ cervical cancer, prostate cancer, or other in-situ cancers
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening and at each tumor assessment), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study intervention
* Has severe hypersensitivity (>= grade 3) to pembrolizumab/BO-112 and/or any of its excipients
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection (HIV 1/2 antibodies). Note: No HIV testing is required unless mandated by local health authority
* Has a known history of active TB (Bacillus tuberculosis)
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator, including dialysis
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment
* Has had an allogenic tissue/solid organ transplant
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guerin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist) are live attenuated vaccines and are not allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-13 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 4 years
  ORR is defined as the proportion of the subjects in the analysis population who have a complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. ORR will be estimated and 95% Clopper-Pearson exact confidence intervals (CIs) will be provided.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From Cycle 1 day 1 (each cycle is 21 days) to the first documented disease progression or death due to any cause, whichever occurs first, assessed up to 4 years]
  Progression will be assessed per RECIST 1.1. PFS will be summarized using the Kaplan Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum).
Time to progression (TTP) | From Cycle 1 day 1 (each cycle is 21 days) to the first documented disease progression, assessed up to 4 years]
  TTP will be summarized using the Kaplan Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum).
Disease control rate (DCR) | Up to 4 years
  DCR is defined as the proportion of subjects who have achieved CR, PR, or stable disease after >= 5 weeks (the start of the window for the first scheduled scan) based on assessments by the site per RECIST 1.1.
Overall survival (OS) | From Cycle 1 day 1 (each cycle is 21 days) to death due to any cause, assessed up to 4 years]
  OS will be summarized using the Kaplan Meier method as well as descriptively (mean, standard deviation, median, first and third quartiles, minimum, maximum). Figures showing the Kaplan-Meier estimates will also be presented. 12-month survival rate will be recorded.
Incidence of adverse events | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Finn, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States